CLINICAL TRIAL: NCT04132986
Title: Multicenter Descriptive Study of Absorbable Biosynthetic Meshes in Contaminated Ventral Hernia Repair
Brief Title: Study of Absorbable Biosynthetic Meshes in Contaminated Ventral Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7398
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Ventral Hernia Repair
Keywords: Ventral hernia repair; Contaminated surgery; Biosynthetic absorbable mesh; Descriptive study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The potential value of biological and biosynthetic meshes is their ability to integrate and remodel the wall in a contaminated environment in complex surgical situations. However, postoperative morbidity and recurrence rate for biologic prostheses are high. The delay to evaluate biosynthetic prostheses is not enough at present, and the high cost of biological prostheses requires a parsimonious use of this type of material. The interest of absorbable biosynthetic prostheses remains to be demonstrated in terms of postoperative complications and long-term recurrence. Current studies have been done on groups with few subjects and in clean surgery.

The primary purpose is to describe the number of complications of the operative site at 12 months, including infectious and noninfectious complications as hematoma and seroma type. The secondary purpose is to describe the number of recurrent ventral hernia at 12 months.

The ventral hernia repair is a frequent operation of general surgery. Thanks to this descriptive work considering the new therapeutic offer with absorbable polymers, it would make possible to update the knowledge of the surgeons and to bring new elements of discussion in the surgical decision.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient ( ≥18 years)
* Patient who has agreed to the use of his medical data for the purposes of this research,
* Patient having been operated between May 2016 and September 2018 in a programmed or urgent surgery, as part of clean / contaminated to dirty surgery at mVHWG grade 3 in the centers participating in the study,
* Patient who benefited between May 2016 and September 2018 from a biosynthetic mesh

Exclusion Criteria:

* Patient who has not consented to the use of her medical data for the purposes of this research,
* Patients who have benefited from the placement of a Phasix® ST biosynthetic mesh in intraperitoneal or Phasix® in retro-muscular prophylaxis,
* Patient under safeguard of justice,
* Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adult patient having been operated between May 2016 and September 2018 in a programmed or urgent surgery, as part of clean / contaminated to dirty surgery at mVHWG grade 3 in the centers participating in the study,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The main criterion will be clinical outcomes : complications and recurrence. It will be expressed in terms of complication according to the Clavien-Dindo classification | Files analysed retrospectily from May 1st, 2016 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie générale et digestive, Strasbourg, France

REFERENCES:
- [Derived] Charleux-Muller D, Hurel R, Fabacher T, Brigand C, Rohr S, Manfredelli S, Passot G, Ortega-Deballon P, Dubuisson V, Renard Y, Romain B. Slowly absorbable mesh in contaminated incisional hernia repair: results of a French multicenter study. Hernia. 2021 Aug;25(4):1051-1059. doi: 10.1007/s10029-020-02366-5. Epub 2021 Jan 25. PMID 33492554